CLINICAL TRIAL: NCT06559605
Title: Clinical and Radiographic Evaluation of Bone Gain Using Customized 3D Printed Zirconia Barrier Versus Titanium Mesh in Combined Ridge Defects in The Aesthetic Zone: A Randomized Clinical Trial
Brief Title: Evaluation of Bone Gain Using Customized 3D Zirconia Barrier Versus Titanium Mesh
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amaal Abdel Nasser Said Mohamed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PER 6-3-1.1
Record Dates: First submitted 2024-07-12; First posted 2024-08-19 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Bone Loss, Alveolar
Keywords: zirconia membrane; titanium membrane; combined bone defect
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Masking of the outcome assessor and patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- zirconia barrier (Active Comparator): Zirconia will be used as a barrier material because it has interesting features and, if compared to titanium, it induces a better fibroblast response. It also shows less biofilm adhesion and less inflammatory response. From the pre-operative CBCT a 3D model of the alveolar jaw bone will be created. A 0.4-0.5 mm-thick barrier will then be designed. It will be designed to cover the planned bone graft and extended a few millimeters wider than the graft perimeter.
  Interventions: Procedure: zirconia barrier
- titanium mesh (Placebo Comparator): Titanium mesh in particular, its clinical suitability for GBR procedures is unmatched by other GBR membranes, due to their exceptional volume stability, titanium meshes are indispensable in the management of vertical or large horizontal bone defects. Titanium meshes not only demonstrate high strength and stiffness but also exhibit good plasticity, allowing them to be perfectly adapted to various bone defects through bending and shaping. Due to titanium mesh's stiffness and sharp edges from cutting and bending, mucosal flaps may be adversely stimulated, leading to mucosal rupture and subsequent mesh exposure
  Interventions: Procedure: titanium mesh

INTERVENTIONS:
Procedure: zirconia barrier — barrier membrane used for guided bone regeneration and augmentation of ridge defect
  Other Names: zirconia membrane
  Arms: zirconia barrier
Procedure: titanium mesh — barrier membrane used for guided bone regeneration
  Arms: titanium mesh

SUMMARY:
Evaluation of clinical and radiographical amount of bone gained using customized 3D printed zirconia barrier compared to titanium mesh in combined ridge defect at the esthetic zone.

DETAILED DESCRIPTION:
After a tooth is extracted, the alveolar process undergoes an inevitable dimensional change as part of the post extraction remodeling process. The alveolar process is reduced both in the vertical and the horizontal dimension. Therefore, Bone augmentation procedures have been employed to address this issue. A number of bone grafting materials and membranes have been used including resorbable and non-resorbable membranes. It is well-established that non-resorbable membranes produce greater bone augmentation than resorbable ones in terms of their ability to generate new bone. However, their complications make them a less popular option in everyday clinical practice.

Zirconia surfaces show prominent osteo-conductivity, also it has low affinity to bacterial plaque, small amounts of inflammatory infiltrate and good soft-tissue integration. Therefore, this study aims to introduce customized-3D zirconia barriers as a predictable alternative to titanium mesh with horizontal bone gain used as primary outcome.

A randomized clinical trial designed to evaluate the amount of bone gained clinically and radiographically using customized 3D printed zirconia barrier compared to titanium mesh with 26 sites with combined ridge defect total sample size, 13 sites per arm. Once patient preparation is completed and the radiographs are acquired, the patient will be assigned into an arm in the study to allow for barrier manufacturing.

For the zirconia group from the pre-operative CBCT a 3D model of the alveolar jawbone will be created. A 0.4-0.5 mm-thick barrier will then be designed. It will be designed to cover the planned bone graft and extended a few millimeters wider than the graft perimeter. The barrier will be milled and sintered, after milling and finishing, the zirconia meshes will be cleaned, dis-infected and sterilized. At the time of the surgery and after administration of anesthesia, the full thickness flap of the atrophic area will be elevated adjacent to the defect site. Autogenous bone particulate will be harvested. Autogenous bone will be harvested by using an auto-chip maker (ACM) bur, autogenous bone chips that collected with ACM bur will be mixed with a xenograft at 50:50 ratio. A try-in of the barrier will be performed before grafting the area to verify whether its adaptation to the recipient site will be correct. A part of the graft will be placed into the atrophic area and the other part of it was placed into the inner side of the barrier. The barrier will be then placed and according to the clinical situation, two or three fixation screws were tightened at 10 N/cm.

The titanium mesh group, an aluminum foil will be adapted to the defect site and used as a guide for trimming the titanium mesh and ensure its adequate fit. The titanium mesh will be polished to prevent dehiscence or premature exposure. It will then stabilize over the particulate graft by 2 mm titanium mini screws at the labial and palatal sides. Releasing incisions of the flaps will be the next step in the procedure. Then, suturing was performed with single and horizontal mattress sutures.

The patient will be instructed to take antibiotics, antiseptic mouth rinse, anti-inflammatory drugs and instructed to apply an ice pack to the treated area for the first 24 hours and to avoid any brushing or trauma to the surgical site for one week.

After 6 months of a healing period a post-operative CBCT will be performed to assess the effectiveness of the GBR procedure, and then Dental implants will be placed according to the bone dimensions. The osteotomy will be initially done using a 4 mm-diameter trephine bur, instead of the pilot drill to acquire a core biopsy. Sequential drilling will then take place until the correct osteotomy size is created for the implant size

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-70 years.
* Bone width less than 4mm
* Vertical bone height less than 9mm
* Periodontally sound neighboring teeth
* Patients with sound vertical occlusal bite dimension
* Good oral hygiene (full mouth plaque control record [PCR] < 25%,full mouth bleeding on probing (BOP) < 25% .
* Patients demonstrating understanding and commitment to the post-operative care regime and the study follow up timeline.
* Good general health (including participants with well-controlled systemic disease)

Exclusion Criteria:

1. Pathological lesions (abscess-cyst-acute infection) in the defect site
2. Systemic diseases that would interfere with bone metabolism
3. Uncontrolled diabetic patients
4. Ongoing treatment or a history of recent chemotherapy or radiotherapy
5. Poor oral hygiene after hygienic phase (Plaque control record over 30%) or Active periodontal disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2026-05-22 (Estimated); Study Completion 2026-11-22 (Estimated)

PRIMARY OUTCOMES:
horizontal bone gain | 6 months
  Horizontal bone gain will be assessed on CBCT after 6 months of bone augmentation

SECONDARY OUTCOMES:
Vertical bone gain | 6 months after barrier placement
  measured on CBCT in a linear dimension as a different in measurement between pre and post operative CBCT.
Quality of bone | 6 months after barrier placement
  The core biopsies will be sectioned and stained with H&E stain for examination under a light microscope. Bone volume will be measured for each specimen and the mean volume for native bone and newly formed bone will be calculated for statistics
Incidence of membrane exposure | up to 4 weeks
  Healing complications including membrane exposure during the period of barrier placement will be recorded and it's evaluated by visual inspection
Membrane exposure area/percentage | up to 4 weeks
  The exposed area will be measured will be assessed by UNC-15 periodontal probe.
Soft tissue thickness | 6 months after barrier placement
  An endodontic spreader with a rubber stopper will be positioned on the soft tissue to record the thickness of the soft tissue.
Procedural time | during the surgery
  Procedural time will be calculated with a stopwatch to measure the time of each procedure and detect differences in the time spend placing and removing the different membranes.
Patient pain | first 12 days after the surgery
  Readings will be recorded by the patient for the first 12 days after the surgery using the visual analogue scale (VAS) which is a descriptive numerical rating scale of 0 to 10.
  0 = No pain 1-3= Mild pain 4-6 = Moderate pain (bearable) 7-10 = Severe pain (unbearable)
Patient satisfaction | 6 months
  Patient will answer questionnaire related to postsurgical and outcome satisfaction (numerical)

CONTACTS AND LOCATIONS:
Overall Officials: Hani El Nahass, Study Director — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt